CLINICAL TRIAL: NCT05984446
Title: Targeting Default Mode Network Dysfunction in Persons At Risk of Alzheimer's Disease with Non-invasive Techniques
Acronym: NEST4AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Michela Pievani, Head, Lab Alzheimer's Neuroimaging & Epidemiology, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GR-2018-12368250
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Default mode network; APOE; rTMS; connectivity
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- real-rTMS (Experimental): 4 daily 25-minutes high-frequency rTMS sessions over one week
  Interventions: Device: real-rTMS
- sham-rTMS (Sham Comparator): 4 daily 25-minutes sham-rTMS sessions over one week
  Interventions: Device: sham-rTMS

INTERVENTIONS:
Device: real-rTMS — Each subject will undergo 4 rTMS sessions using a 70-mm figure-eight coil (20Hz for 25 minutes). Target localization will be performed with a stereotaxic neuronavigation system.
  Arms: real-rTMS
Device: sham-rTMS — The sham condition will match the real-rTMS protocol, but a sham coil will be used.
  Arms: sham-rTMS

SUMMARY:
Default mode network (DMN) dysfunction is a well-established feature of Alzheimer's Disease (AD) and is already present in preclinical stages and in subjects at risk for AD, thus offering a potential target for early intervention. Non-invasive stimulation techniques are candidate approaches to modulate network dysfunction, however interventions specifically targeting subjects at risk for AD are lacking. This project will test a non-invasive intervention to modulate the DMN in cognitively healthy older adults carrying the main genetic risk factor for AD, the APOE e4 allele. The proposal will non-invasively stimulate the DMN in at risk subjects and will assess the neuronal-cognitive effect of this approach with multimodal neuroimaging and neurophysiological techniques.

DETAILED DESCRIPTION:
Sixty-four participants will be enrolled (n=32 APOE e4 carriers, 32 non-carriers as reference group) and will undergo rTMS stimulation, TMS with concurrent electroencephalography (TMS-EEG), multimodal imaging (resting-state and task functional MRI, and diffusion tensor imaging) and cognitive assessment at baseline, after the intervention (week 1) and after 2 months. Participants will be randomized to 2 groups: active DMN stimulation (real-rTMS) or placebo (sham-rTMS). Each subject will undergo a rs-fMRI scan before the intervention to derive individualized DMN stimulation targets. rTMS will be applied over the left inferior parietal lobule node of the DMN.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60 years and older
* MMSE score > 24

Exclusion Criteria:

* Pathological scores in at least two standardized cognitive tests
* Participation in other interventional studies
* Known carriers of an autosomal dominant genetic mutation associated to AD
* Neurological, psychiatric or medical conditions not compatible with the study

Exclusion Criteria for MRI and rTMS:

* metal implants, pace-makers, prosthetic heart valves
* claustrophobia
* history of epilepsy
* pregnancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Change in DMN connectivity on rs-fMRI following real-rTMS compared to sham-rTMS in APOE4 carriers | Baseline, post rTMS (1 week)
  Default mode network (DMN) mean functional connectivity is assessed on resting state functional MRI. Higher values denote greater functional connectivity. A positive change at post rTMS compared to baseline represents an increase in resting-state functional connectivity.
Change in DMN connectivity on TMS-EEG following real-rTMS compared to sham-rTMS in APOE4 carriers | Baseline, post rTMS (1 week)
  Single pulse TMS will be applied with concurrent EEG to derive online measures of cortical excitability and connectivity. The response in the natural frequency of the target area will index cortical excitability. Effective connectivity will be measured through amplitude and latency of TEPs.

SECONDARY OUTCOMES:
Change in task-fMRI associative memory performance following real-rTMS compared to sham-rTMS in APOE4 carriers | Baseline, post rTMS (1 week)
  Memory is assessed on task fMRI using a face-name associative paradigm

OTHER OUTCOMES:
Change in DMN connectivity on rs-fMRI following real-rTMS in APOE4 carriers compared to non-carriers | Baseline, post rTMS (1 week)
  Default mode network (DMN) mean functional connectivity is assessed on resting state functional MRI. Higher values denote greater functional connectivity. A positive change at post rTMS compared to baseline represents an increase in resting-state functional connectivity.
Change in DMN connectivity on TMS-EEG following real-rTMS in APOE4 carriers compared to non-carriers | Baseline, post rTMS (1 week)
  Single pulse TMS will be applied with concurrent EEG to derive online measures of cortical excitability and connectivity. The response in the natural frequency of the target area will index cortical excitability. Effective connectivity will be measured through amplitude and latency of TEPs.
Change in task-fMRI associative memory performance following real-rTMS in APOE4 carriers compared to non-carriers | Baseline, post rTMS (1 week)
  Memory is assessed on task fMRI using a face-name associative paradigm
Change in cognition following real-rTMS in APOE4 carriers compared to non-carriers | Baseline, post rTMS (1 week)
  Cognition is assessed with the MMSE, the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), the Free and Cued Selective Reminding Test (FCSRT), and the preclinical Alzheimer cognitive composite (PACC) score.
Change in cognition following real-rTMS compared to sham-rTMS in APOE4 carriers | Baseline, post rTMS (1 week)
  Cognition is assessed with the MMSE, the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), the Free and Cued Selective Reminding Test (FCSRT), and the preclinical Alzheimer cognitive composite (PACC) score.
Change in cognition following real-rTMS compared to sham-rTMS in APOE4 carriers | Baseline, post rTMS (2 months)
  Cognition is assessed with the MMSE, the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), the Free and Cued Selective Reminding Test (FCSRT), and the preclinical Alzheimer cognitive composite (PACC) score.

CONTACTS AND LOCATIONS:
Overall Officials: Michela Pievani, Principal Investigator — IRCCS Centro San Giovanni di Dio Fatebenefratelli
Locations (1):
- IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pievani M, Mega A, Quattrini G, Guidali G, Ferrari C, Cattaneo A, D'Aprile I, Mascaro L, Gasparotti R, Corbo D, Brignani D, Bortoletto M. Targeting Default Mode Network Dysfunction in Persons at Risk of Alzheimer's Disease with Transcranial Magnetic Stimulation (NEST4AD): Rationale and Study Design. J Alzheimers Dis. 2021;83(4):1877-1889. doi: 10.3233/JAD-210659. PMID 34459405
- [Background] Bagattini C, Brignani D, Bonni S, Quattrini G, Gasparotti R, Pievani M. Functional Imaging to Guide Network-Based TMS Treatments: Toward a Tailored Medicine Approach in Alzheimer's Disease. Front Neurosci. 2021 Jul 5;15:687493. doi: 10.3389/fnins.2021.687493. eCollection 2021. PMID 34290585